CLINICAL TRIAL: NCT02367599
Title: Effect of Vitamin D Supplementation on Bone Turnover Markers During Tenofovir-Emtricitibine Pre-Exposure Prophylaxis in Men Who Have Sex With Men; A Sub-study of CCTG 595
Brief Title: Effect of Vitamin D Supplementation on Bone Turnover Markers During PrEP in MSM
Acronym: CCTG595VitD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Southern California (Other); University of California, Los Angeles (Other); City of Long Beach Department of Health and Human Services (Other Government); California HIV/AIDS Research Program (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCTG 595 Vitamin D Sub-Study
Record Dates: First submitted 2015-02-10; First posted 2015-02-20 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Patient Adherence
Keywords: PrEP; Pre exposure Prophylaxis; Truvada; CCTG; 595; Vitamin D; Bone mineral density
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Supplement + PrEP (Active Comparator): Subjects enrolled into this sub-study will be provided Vitamin D 4000IU/day for 24 Weeks in addition to their PrEP provided through the main study.
  Interventions: Drug: Vitamin D Supplement
- PrEP Only (No Intervention): Subjects not enrolled into this sub-study will continue receiving PrEP through the main study. Subjects taking unsupplemented PrEP may still be used as matched controls to sub-study subjects.

INTERVENTIONS:
Drug: Vitamin D Supplement — Subjects enrolled into this sub-study will be provided Vitamin D 4000IU/day for 24 Weeks.
  Arms: Vitamin D Supplement + PrEP

SUMMARY:
CCTG 595 is an open-label clinical trial of the effect of a text messaging intervention vs. standard of care on adherence to Truvada as PrEP in MSM at increased risk for HIV infection (ClinicalTrials.gov Identifier: NCT01761643). Eligible subjects for this matched case control substudy will receive vitamin D 4000 IU/day for 24 weeks, from week 24 through week 48. In CCTG 595, plasma from participants are being collected and stored at entry and every 12 weeks. These plasma samples will be used to measure P1NP, CTX, PTH, and vitamin D levels in both cases and controls at entry, week 24, and week 48.

DETAILED DESCRIPTION:
A total of 50 HIV-uninfected men who have sex with men (MSM) and male to female (M to F) transgender individuals already enrolled in CCTG 595 will be offered participation in the sub-study at Week 24 of the main study. All subjects enrolled into the sub-study will be provided Vitamin D 4000 IU/day supplements in addition to their PrEP at Weeks 24 and 36; clinic visits will proceed normally per main study protocol. Upon completion of the sub-study subjects will continue on the main study.

The primary endpoint, bone turnover markers, will be measured from Week 24 to Week 48 via plasma samples collected through the main study. Concurrent controls who are not enrolled in the vitamin D substudy who are reporting supplementation with < 400 IU of vitamin D/day will be matched 1:1 by randomization arm in the CCTG 595 main study (text messaging arm vs. standard of care), age (± 5 years), race/ethnicity, season of study entry, and BMI (± 3 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet CCTG 595 inclusion criteria.

Exclusion Criteria:

* All subjects must meet CCTG 595 exclusion criteria.
* Current or prior use of bisphosphonate therapy.
* Current use of Vitamin D supplements greater than 400 IU/day.
* Current use of androgenic hormones or growth hormones.
* History of nephrolithiasis (kidney stones).
* History of fragility fracture.
* No use of tenofovir prior to entry into CCTG 595

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Dube, MD, Study Chair — CCTG, USC; Sheldon Morris, MD, Principal Investigator — UC San Diego AntiViral Research Center (AVRC)
Locations (3):
- United States (3):
  - University Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the parent trial (CCTG 595) were offered the opportunity to enroll in this sub-study providing Vitamin D supplementation to HIV pre-exposure prophylaxis (PrEP).
Pre-assignment Details: 48 enrolled, 48 matched from parent study. Total 96 evaluated participants.
Groups:
- Vitamin D Supplement + PrEP: Subjects enrolled into this sub-study will be provided Vitamin D 4000IU/day for 24 weeks in addition to their PrEP provided through the parent trial.
- PrEP Only Matched Group: A cohort of parent trial participants will be selected to match subjects enrolled in the sub-study to serve as comparative controls.
Period: Overall Study
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PrEP Only Matched Group: A cohort of main-study participants will be selected to match subjects enrolled in the sub-study to serve as controls for comparison.
- Total: Total of all reporting groups
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.5 [28 to 37.5] | 33.0 [29 to 38.5] | 33.2 [28.5 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 48 | 48 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 25 | 51
  Black | 13 | 14 | 27
  Asian | 2 | 2 | 4
  Multiracial | 6 | 6 | 12
  Hispanic | 16 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Procollagen Type 1 N-terminal Propeptide (a Marker of Bone Formation) [P1NP] Levels
Description: To compare the change in P1NP levels from Week 24 through Week 48 among subjects (cases) who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls
Time Frame: Weeks 24-48
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
Number analyzed (Participants) | 48 | 48
pg/mL | -27.6 (49.9) | -2.5 (40.2)

2. Secondary Outcome: Change in CTX-1 Levels
Description: To compare the change in CTX-1 levels from Week 24 through Week 48 among subjects (cases) who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls
Time Frame: Weeks 24-48
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
Number analyzed (Participants) | 48 | 48
ng/mL | 0.03 (1.12) | 0.29 (2.10)

3. Secondary Outcome: Change in PTH Levels
Description: To compare the change in PTH levels from Week 24 through Week 48 among subjects (cases) who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls
Time Frame: Weeks 24-48
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
Number analyzed (Participants) | 48 | 48
pg/mL | 57.3 (128.9) | 108.4 (210.5)

4. Secondary Outcome: Change in 25-OH Vitamin D3 Levels
Description: To compare the change in 25-OH vitamin D3 levels from Week 24 through Week 48 among subjects (cases) who receive vitamin D 4000 IU/day to the change in levels seen in matched unsupplemented controls
Time Frame: Weeks 24-48
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
Number analyzed (Participants) | 48 | 48
ng/mL | 4.4 (16.2) | -0.9 (13.7)

ADVERSE EVENTS:
Time Frame: Weeks 24-48
Arm/Group | Vitamin D Supplement + PrEP | PrEP Only Matched Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02367599/Prot_SAP_000.pdf